CLINICAL TRIAL: NCT06901349
Title: A Phase 2b Double-Blind, Randomized, Placebo-Controlled Study of Bimagrumab and Tirzepatide, Alone or in Combination, to Investigate the Efficacy and Safety in Adult Participants With Obesity or Overweight With Type 2 Diabetes
Brief Title: A Study of Bimagrumab (LY3985863) and Tirzepatide (LY3298176), Alone or in Combination, in Participants With Obesity or Overweight With Type 2 Diabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated for strategic business reasons
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27328; J4Z-MC-GIDI (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-03-24; First posted 2025-03-28 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Overweight
Keywords: Type 2 Diabetes; Muscle; Lean; Fat
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2; Platelet Glycoprotein IV Deficiency | interventions — bimagrumab; Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Bimagrumab Dose 1 + Tirzepatide Placebo (Experimental): Participants will receive bimagrumab subcutaneously (SC) and tirzepatide placebo SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide Placebo
- Bimagrumab Dose 2 + Tirzepatide Placebo (Experimental): Participants will receive bimagrumab SC and tirzepatide placebo SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide Placebo
- Tirzepatide Dose 1 + Bimagrumab Placebo (Experimental): Participants will receive tirzepatide SC and bimagrumab placebo SC
  Interventions: Drug: Tirzepatide; Drug: Bimagrumab Placebo
- Tirzepatide Dose 2 + Bimagrumab Placebo (Experimental): Participants will receive tirzepatide SC and bimagrumab placebo SC
  Interventions: Drug: Tirzepatide; Drug: Bimagrumab Placebo
- Bimagrumab Dose 2 + Tirzepatide Dose 1 (Experimental): Participants will receive bimagrumab SC and tirzepatide SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide
- Bimagrumab Dose 1 + Tirzepatide Dose 1 (Experimental): Participants will receive bimagrumab SC and tirzepatide SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide
- Bimagrumab Dose 2 + Tirzepatide Dose 2 (Experimental): Participants will receive bimagrumab SC and tirzepatide SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide
- Bimagrumab Dose 1 + Tirzepatide Dose 2 (Experimental): Participants will receive bimagrumab SC and tirzepatide SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide
- Bimagrumab Placebo + Tirzepatide Placebo (Placebo Comparator): Participants will receive bimagrumab placebo SC and tirzepatide placebo SC
  Interventions: Drug: Bimagrumab Placebo; Drug: Tirzepatide Placebo

INTERVENTIONS:
Drug: Bimagrumab — Administered SC
  Other Names: LY3985863
  Arms: Bimagrumab Dose 1 + Tirzepatide Dose 1; Bimagrumab Dose 1 + Tirzepatide Dose 2; Bimagrumab Dose 1 + Tirzepatide Placebo; Bimagrumab Dose 2 + Tirzepatide Dose 1; Bimagrumab Dose 2 + Tirzepatide Dose 2; Bimagrumab Dose 2 + Tirzepatide Placebo
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Bimagrumab Dose 1 + Tirzepatide Dose 1; Bimagrumab Dose 1 + Tirzepatide Dose 2; Bimagrumab Dose 2 + Tirzepatide Dose 1; Bimagrumab Dose 2 + Tirzepatide Dose 2; Tirzepatide Dose 1 + Bimagrumab Placebo; Tirzepatide Dose 2 + Bimagrumab Placebo
Drug: Bimagrumab Placebo — Administered SC
  Arms: Bimagrumab Placebo + Tirzepatide Placebo; Tirzepatide Dose 1 + Bimagrumab Placebo; Tirzepatide Dose 2 + Bimagrumab Placebo
Drug: Tirzepatide Placebo — Administered SC
  Arms: Bimagrumab Dose 1 + Tirzepatide Placebo; Bimagrumab Dose 2 + Tirzepatide Placebo; Bimagrumab Placebo + Tirzepatide Placebo

SUMMARY:
The main purpose of this study is to see how well and how safely bimagrumab, tirzepatide, and the combination, work in lowering body weight in participants with obesity or overweight and type 2 diabetes. Participation in the study will last about 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes
* Have a BMI of ≥27 kilograms per square meter (kg/m2)
* Have had a stable body weight for the 3 months prior to randomization (<5% body weight gain and/or loss)

Exclusion Criteria:

* Have a prior or planned surgical treatment for obesity,
* Have type 1 diabetes, latent autoimmune diabetes, or history of ketoacidosis or hyperosmolar state or coma
* Have poorly controlled hypertension
* Have any of the following cardiovascular conditions within 3 months prior to screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * unstable angina, or
  * hospitalization due to congestive heart failure
* Have a history of New York Heart Association (NYHA) Functional Classification III or IV congestive heart failure
* Have ongoing or a history of frequent intermittent or chronic tachyarrhythmia syndromes
* Have ongoing or a history of bradyarrhythmias other than sinus bradycardia
* Have renal impairment
* Have a history of symptomatic gallbladder disease within the past 2 years
* Have signs and symptoms of any liver disease
* Have a disease or condition known to cause gastrointestinal malabsorption or a known clinically significant gastric emptying abnormality
* Have a history of acute or chronic pancreatitis
* Currently taking or have taken medications that may cause significant weight gain or promote weight loss within 3 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 36

SECONDARY OUTCOMES:
Percent Change from Baseline in Total Body Fat Mass by Dual-Energy X-Ray Absorptiometry (DXA) | Baseline, Week 36
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 36
Percentage of Participants Achieving ≥5% Body Weight Reduction | Baseline, Week 36
Percentage of Participants Achieving ≥10% Body Weight Reduction | Baseline, Week 36
Percentage of Participants Achieving ≥15% Body Weight Reduction | Baseline, Week 36
Change from Baseline in Waist Circumference | Baseline, Week 36
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 36
Change from Baseline in Waist-to-Height Ratio (WHtR) | Baseline, Week 36
Percent Change from Baseline in Visceral Adipose Tissue (VAT) by Magnetic Resonance Imaging (MRI) | Baseline, Week 36
Change from Baseline in Liver Fat by MRI | Baseline, Week 36
Percent Change from Baseline in High-Sensitivity C-Reactive Protein (hsCRP) | Baseline, Week 36
Percent Change from Baseline in Total Cholesterol | Baseline, Week 36
Percent Change from Baseline in Triglycerides (TG) | Baseline, Week 36
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 36
Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve (AUC-ss) of Bimagrumab | Predose through Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (50):
- United States (25):
  - Yuma Clinical Trials, Yuma, Arizona
  - Orange County Research Center, Lake Forest, California
  - Healthy Brain Clinic, Long Beach, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - Global Health Research Center, Inc., Miami Lakes, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Balanced Life Health Care Solutions/SKYCRNG, Lawrenceville, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - Family First Medical Center, Idaho Falls, Idaho
  - Deaconess Clinic- Gateway, Newburgh, Indiana
  - Kur Research - Columbia Medical, Columbia, Maryland
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Remington-Davis, Inc, Columbus, Ohio
  - Central States Research, Tulsa, Oklahoma
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Activian Clinical Research, Kingwood, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Argentina (4):
  - CIPREC, Buenos Aires, Buenos Aires F.D.
  - Centro Médico Viamonte, Buenos Aires, Buenos Aires F.D.
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires, Buenos Aires F.D.
  - CIPREC, Buenos Aires
- Canada (7):
  - Richmond Clinical Trials, Richmond, British Columbia
  - Centricity Research Brampton Endocrinology, Brampton, Ontario
  - Premier Clinical Trial Network, Hamilton, Ontario
  - Your Research Network, Niagara Falls, Ontario
  - Centricity Research Pointe-Claire Multispecialty, Pointe-Claire, Quebec
  - Diex Recherche Trois-Rivieres, Trois-Rivières, Quebec
  - Diex Recherche Quebec, Québec
- China (6):
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi, Henan
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
- Japan (8):
  - Tokuyama Clinic, Mihama-ku,Chiba City, Chiba
  - Hayashi Diabetes Internal Medicine Clinic, Chigasaki, Kanagawa
  - Shonan Takai Clinic, Kamakura, Kanagawa
  - Takai Internal Medicine Clinic, Kamakura-shi, Kanagawa
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - The Institute of Medical Science, Asahi Life Foundation, Chuo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Bimagrumab (LY3985863) and Tirzepatide (LY3298176), Alone or in Combination, in Participants with Obesity or Overweight with Type 2 Diabetes — https://trials.lilly.com/en-US/trial/587595